# **Evaluation of the Effects of Silk and Polyester Suture on Postoperative Complications in Lower**

# **Impacted Third Molar Teeth Surgery**

Levent Ciğerim DDS, PhD <sup>1</sup>, Mehmet Güzel <sup>1</sup>, Abdulrahman Alghalaeini <sup>1</sup>, Zeynep Dilan Orhan <sup>1</sup> Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery, Van,

**TURKEY** 

Corresponding author: Levent Ciğerim

Address: Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery,

Van, Turkey Postal Code: 65080

E-mail address: <u>levent139@hotmail.com</u> Phone:+905321633287 Office Phone: 904322251744 Fax:

+904322251747

#### Levent CİĞERİM

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery levent139@hotmailmail.com,
+905321633287, <a href="https://orcid.org/0000-0001-5218-8568">https://orcid.org/0000-0001-5218-8568</a>

#### Mehmet GÜZEL

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <a href="mailto:dtmehmetguzel@gmail.com">dtmehmetguzel@gmail.com</a>, +905363609854, <a href="https://orcid.org/0000-0002-9621-0496">https://orcid.org/0000-0002-9621-0496</a>

### Abdulrahman Alghalaeini

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <u>dentist.a.gh@gmail.com</u>, +905355524762, <a href="https://orcid.org/0000-0002-0443-5592">https://orcid.org/0000-0002-0443-5592</a>

#### Zeynep Dilan Orhan

Van Yuzuncu Yil University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery <a href="mailto:zeynepdilanorhan@gmail.com">zeynepdilanorhan@gmail.com</a>, +905425525525, <a href="https://orcid.org/0000-0003-1333-9073">https://orcid.org/0000-0003-1333-9073</a>

# VAN YÜZÜNCÜ YIL UNIVERSITY DURSUN ODABAŞ MEDICAL CENTER INFORMED CONSENT FORM FOR RESEARCH

## Dear patient,

Please read this document carefully and listen carefully to what we have said. Detailed information about the research; Detailed information about your rights, benefits and risks of the research can be found in this document. The purpose of these statements is to inform you about your health. Please indicate what you do not understand, your questions will be explained in detail. You can leave the research at any stage of the research if you think that your questions are not adequately explained after you accept to participate in the research or for any other reason. During the research period, the health problems arising from our research will be treated in our hospital immediately. You will not be charged an additional fee for participating in this research, nor will you be paid. Thank you for participating in our research.

**Name of the Study:** Evaluation of the Effects of Silk and Polyester Suture on Postoperative Complications in Lower Impacted Wisdom Teeth Surgery

The subject, purpose, method, time and process to be used of the research: Our research is about the postoperative success of sutures placed after tooth extraction. It is aimed to determine which material is effective in the simple suture technique.

Suggested action/process for research: More effective wound closure methods with fewer complications have positive effects on postoperative recovery. Suturing is the most commonly used wound closure technique after lower impacted wisdom tooth surgery. Suturing, which is the last step of the operation, contributes to wound healing in order to reposition and stabilize the tissue components and to control bleeding. In our study, it was aimed to evaluate the efficacy of silk and polyester sutures used in wound closure techniques, which are frequently used in lower impacted wisdom teeth surgery. The study was carried out on 30 patients who applied to Van Yüzüncü Yıl University, Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery, Silk suture will be used on one side of the patients and polyester suture will be used on the other side. Sutures with a diameter of 3/8 and a thickness of 4/0 with reverse sharp needles were used in the groups. When the patients first applied to the clinic, their anamnesis was taken and panoramic images were taken after clinical evaluations were made. In this randomized, single-blind, split-mouth study, evaluations were made with preoperative face measurements (for evaluation of swelling), maximum mouth opening (for evaluation of trismus) and periodontal measurements for all patients. The mentioned measurements and evaluations were repeated on the 2nd and 7th postoperative days. In addition, postoperative pain was evaluated with the VAS scale, which the patients would fill in themselves. The same surgical procedure will be performed by the same surgeon for all patients. After local anesthesia (80 mg Articaine hydrochloride + 0.02mg Epinephrine bitartrate, 2ml Maxicain Fort), a 3-corner flap containing the vertical incision passing through the mesial of the number 7 was lifted, the bone would be removed under saline cooling and the teeth were separated when necessary. Afterwards, the extraction sockets will be irrigated with saline to control bleeding, and the area is closed primarily with silk or polyester suture material.

All patients received postoperative analgesics (1200mg Ibuprofen daily, BRUFEN 600mg Film Tablet 2\*1) and antiseptic mouthwash (0.15% Benzydamine hydrochloride and 0.12% Chlorhexidine gluconate, 200 ml Andorex Gargara 3\*1).

Data were collected and evaluated statistically.

Study-specific risks during the study: Allergic reaction

**Possible benefits of the research:** The effectiveness of prf and i-prf-impregnated collagen plug on post-operative complications and wound healing will be determined after the impacted third molar tooth surgery.

**Anesthesia:** Mandibular block anesthesia will be performed during the treatment.

| Phone. No: Name surname: Date of birth: Adress: | Name-Surname of the Physician<br>Responsible for the Research:<br>Associate Professor Levent CİĞERİM<br>Institution Registration Number: 5086<br>Signature: |
|---|---|
| History:: | |
| The Participant's and/or Legal Representative to Get Consent in Emergency Situations | |
| 1. I was invited to the research after I received the preliminary information about the research explained in a clear and simple way and after reading the consent form in my hand. subject invitation; I agreed. 1 did not accept. 2. I have read and listened to the points to be considered in the research. I asked my questions about the research. Required enlightening answers I got it. 1 didn't get it, I don't understand. 3. Provided that my identity is kept confidential and used only for educational and research purposes, I may be photographed during the intervention/treatment to be applied to me, that my data can be used retrospectively or recorded. I allow 1 do not allow. 4. I learned the benefits and possible risks of diagnostic interventions, medical and surgical treatments, and the procedures to be done. I agree. 1 do not accept. 5. Since I can't read/write the research information process or I don't want to decide on my own joined. 6. The data received by me regarding the research will be kept confidential, i know i don't know 7. I have the right to withdraw from the research at any time, i know i don't know 8. I will not charge/pay any fee as a result of the research; i know i don't know 9. If a medical risk arises, free medical treatment will be provided. i know i don't know 12. When I encounter a health problem during the research; at any hour, Dt. I know that I can call Mehmet GÜZEL at 05363609854 (mobile) and at YYU Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery. | |
| Dear patient/ participant/, please read the following articles carefully and fill in the relevant blank or tick the relevant box | |
| <b>Funding of the research:</b> You will not be charged an additional fee for participating in this research and you will not be paid any money. | |
| Anesthesia: Mandibular block anesthesia will be performed during the treatment. | |